CLINICAL TRIAL: NCT04588688
Title: Mifepristone Dynamic Testing for Diagnosis for Central Adrenal Insufficiency
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: low recruitment
Sponsor: Tobias Else (Other)
Collaborators: Corcept Therapeutics (Industry)
Responsible Party: Sponsor-Investigator, Tobias Else, Assistant Professor, Department of Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HUM00160641
Record Dates: First submitted 2020-10-09; First posted 2020-10-19 (Actual); Results first posted 2023-06-12 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-05

CONDITIONS: Central Adrenal Insufficiency; Mifepristone
Keywords: Insulin Tolerance Test
MeSH Terms: interventions — Mifepristone

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Mifepristone (Experimental): Patients will be provided a single dose of 600 milligram (mg) mifepristone to be administered orally, and subjects will be instructed to take the drug between 10PM and 11PM on Day 1.
  Interventions: Drug: Mifepristone

INTERVENTIONS:
Drug: Mifepristone — Mifepristone is a selective antagonist of the progesterone receptor at low doses and blocks the glucocorticoid receptor (GR-II) at higher doses. Mifepristone has high affinity for the GR-II receptor but little affinity for the GR-I (MR, mineralocorticoid) receptor.
  Other Names: KORLYM®, C1073, RU486

SUMMARY:
The researchers propose the use of mifepristone as an alternative way to test for Central Adrenal Insufficiency (CAI). They want to assess the feasibility of recruitment and the efficacy of the purposed method.

DETAILED DESCRIPTION:
Recruitment for this trial was legally opened on February 17, 2020. When the record was first released, it incorrectly listed the recruitment status as "Not Yet Recruiting." This mistake was noticed before the first participant actually enrolled, May 5, 2021. The decision to terminate for low recruitment was made on Sept 7, 2022, approximately 30 months later, as at that point it was deemed impossible to reach the initial enrollment target of 26.

ELIGIBILITY:
Inclusion Criteria (1 of the following):

* Completed insulin tolerance testing (ITT) at University of Michigan from 2012 to present.
* Are scheduled to complete ITT.
* Are clinically suspected to have adrenal insufficiency but have not undergone ITT.

Exclusion Criteria:

* Female patients who are of child-bearing potential (defined as a sexually mature woman who has not undergone hysterectomy, bilateral oophorectomy bilateral salpingectomy or bilateral tubal ligation/occlusion, at least 12 weeks prior to screening, or who has not been naturally postmenopausal for at least 24 consecutive months prior to study enrollment) and not using non-hormonal contraception.
* Female patients not willing to use non-hormonal contraception for one month following treatment.
* Women who are pregnant or breast feeding.
* Patients with an existing diagnosis of adrenal insufficiency who are on any glucocorticoid replacement other than oral hydrocortisone or prednisone.
* Patients on medications that are strong CYP3A
* Patients taking other medications metabolized by CYP3A
* Patients who have a history of QT prolongation and patients with any recent abnormal electrocardiogram (ECG).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2021-05-05 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tobias Else, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: The results from the insulin tolerance test (ITT) served to group the participants into two arms for analysis: high suspicion for adrenal sufficiency (maximum cortisol greater than or equal to 15 microg/dl) or high suspicion for adrenal insufficiency (maximum cortisol less than 15 microg/dl). The ITT serves as the gold standard and the cut-off of 15 microg/dl was used as a conservative cut-off in accordance with local experience with this test.
Period: Overall Study
Arm/Group | Mifepristone
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Greater or Equal to 15 Max Cortisol: Suspected adrenal sufficient by ITT.
- Less Than 15 Max Cortisol: Suspected adrenal insufficient by ITT.
- Total: Total of all reporting groups
Arm/Group | Greater or Equal to 15 Max Cortisol | Less Than 15 Max Cortisol | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Customized [Count of Participants; unit: Participants]
  50 - 59 years | 2 | 0 | 2
  60 - 69 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 0 | 2
  Male | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 0 | 1
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 1 | 3
Peak cortisol measured after Insulin Tolerance Testing (ITT) [Mean (Standard Deviation); unit: micrograms per deciliter] — Peak cortisol measured in participants following ITT. Population: Only 1 participant was in the ITT Less Than 15 Max Cortisol arm. Data are not shared to preserve privacy.
  micrograms per deciliter
    number analyzed (Participants) | 2 | 0 | 2
    (all) | 24.4 (3.15) |  | 24.4 (3.15)

OUTCOME MEASURES:

1. Primary Outcome: Number of Study Participants Recruited
Description: Because this was a feasibility trial, the goal was to see how many participants could be successfully recruited. The original intent was for the recruitment period to be for 36 months, with a target enrollment of 26 participants. The trial opened for recruitment on February 17, 2020. Because of low enrollment, the decision to terminate was made on September 7, 2022, approximately 30 months later.
Time Frame: Up to 88 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone
Number analyzed (Participants) | 3
Participants | 3

2. Primary Outcome: Number of Study Participants With Complete Study Data Captured
Description: Because this was a feasibility trial, the goal was to see how many participants could be successfully recruited. The original intent was for the recruitment period to be for 36 months, with a target enrollment of 26 participants. Because of low enrollment, the decision to terminate was made after the trial had been open for recruitment for approximately 30 months (February 17, 2020 - September 7, 2022).
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Mifepristone
Number analyzed (Participants) | 3
Participants | 3

3. Secondary Outcome: Peak Cortisol Measured After Mifepristone
Description: Serum cortisol was collected the day after mifepristone administration and insulin tolerance test insulin tolerance test (ITT).
Time Frame: Day 2 (day after mifepristone administration)
Population: Only 1 participant was in the ITT Less Than 15 Max Cortisol arm. Results are not shared to preserve privacy.
Measure: Mean (Standard Deviation); unit: micrograms per deciliter
Groups:
- ITT Greater or Equal to 15 Max Cortisol: Suspected adrenal sufficient by ITT.
- ITT Less Than 15 Max Cortisol: Suspected adrenal insufficient by ITT.
Arm/Group | ITT Greater or Equal to 15 Max Cortisol | ITT Less Than 15 Max Cortisol
Number analyzed (Participants) | 2 | 0
micrograms per deciliter | 13.9 (0.75) |

4. Secondary Outcome: Absolute ACTH After Mifepristone
Description: ACTH level 8:00 am (Day 2) following administration of mifepristone the night before at 10:00 pm.
Time Frame: Day 2 (day after mifepristone administration)
Population: Only 1 participant was in the ITT Less Than 15 Max Cortisol arm. Results are not shared to preserve privacy.
Measure: Mean (Standard Deviation); unit: Picogram per milliliter
Arm/Group | Greater or Equal to 15 Max Cortisol | Less Than 15 Max Cortisol
Number analyzed (Participants) | 2 | 0
Picogram per milliliter | 18.5 (1.5) |

ADVERSE EVENTS:
Time Frame: Day 2, Day 7, and Day 30
Arm/Group | Mifepristone
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-18): https://cdn.clinicaltrials.gov/large-docs/88/NCT04588688/Prot_SAP_000.pdf